CLINICAL TRIAL: NCT02862197
Title: Invasive Monitoring of Pulmonary Artery Pressure (PAP) Among Dialysis Treated Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Responsible Party: Principal Investigator, Marjo Soini, study coordinator, Joint Authority for Päijät-Häme Social and Health Care
Other Study IDs: Q298diarnro18/2016
Record Dates: First submitted 2016-03-29; First posted 2016-08-10 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: End Stage Renal Disease; Cardiac Insufficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: hemodialysis treated patients as described in the inclusion of the study

SUMMARY:
The purpose of this study is examine whether invasive pulmonary artery pressure (PAP) monitoring could be beneficial for the patients in dialysis treatment. Ten implantable pressure sensors (CardioMEMS ®) will be implanted and the PAPs of the individual participants are recorded during and in between the routine dialysis treatment sessions. This is an exploratory pilot study, where major interest lies in the values and changes in PAP in relation to other hemodynamic parameters among patients in dialysis treatment. Implanted device is only monitoring the patient without any effect on the actual treatment.

DETAILED DESCRIPTION:
Dialysis treatment is hemodynamically problematic in up to one third of the patients. Particularly, estimation of the adequate fluid removal during the dialysis can be difficult. Removing too much fluid can lead to dehydration, hypotension and dizziness, and insufficient removals can lead to fluid accumulation and worsening of possible heart failure. Both under- and overestimation of the fluid removal have been connected to increased mortality. Balancing the fluid balance is especially challenging in patients with simultaneous heart failure.

Several measures are made and precautions taken during the dialysis to optimize the ultrafiltration individually for each patient. The key question in the estimation of the right amount of ultrafiltration is, how much and at what speed fluid can be safely removed from the patient without critically lowering the filling and preload of the heart.

The results of the CHAMPION trial show that therapy guided by PAP is superior to conventional way in estimating the optimal fluid balance among heart failure patients. Compared to the heart failure patients in the CHAMPION trial, the ESRD patients share some similarities. In both groups, estimating the fluid balance is crucial, but difficult. The changes in fluid balance among ESRD patients are much larger.

In the present study the investigators aim to evaluate the potential of invasive measured PAP in the context of dialysis treatment for patients with end-stage renal disease (ESRD).

After the implantation the basic medical history is taken, echocardiography is made, and their laboratory measurements are recorded. Participants are then monitored during their routine dialysis treatment twice a week over the period of 1 month. In addition twice a day measurement is recorded in home during the study.

PAP measures and its changes are then compared to all the haemodynamical data available including blood volume, systolic and diastolic blood pressure, heart rate, hematocrit measures and bioimpedance measurement during the dialysis treatment.

ELIGIBILITY:
Inclusion Criteria (In addition to details described in "Study Population Description"):

* Subject who is eligible for a CardioMEMS device per physician discretion
* Subject is living at home
* Subject's ability to take part of the study will be discussed with their treating nephrologist.
* Subject is willing and capable of providing informed consent, participating in all associated study activities

Exclusion Criteria:

* Any non-cardiac or non-renal medical condition causing the life-expectancy to be less than one year.
* The patient is not able to take part of the study or the study can be considered to be harmful for the patient in the opinion of the investigator or the treating nephrologist.
* Age >75 years
* Age <18 years
* Probable noncompliance
* Subjects with an active infection
* Subjects who, in the investigator's opinion, are unable to tolerate a right heart catheterization
* Subjects who have had a major cardiovascular event (e.g., myocardial infarction, open heart surgery, stroke, etc.) within 2 months of the baseline visit
* Subjects with a device (Pacemaker/Implantable Cardioverter-Defibrillator/CRT) implanted < 30 days prior to enrollment
* Subjects with congenital heart disease or mechanical right heart valve(s)
* Subjects likely to undergo heart transplantation or ventricular assist device implantation within 6 months of the baseline visit
* Subjects with known coagulation disorders or subjects who are unable to take two types of blood thinning medications or anticoagulation therapy for one month after the sensor is implanted.
* Subject is enrolled in another study with an active treatment arm
* Pregnancy
* Diameter of Pulmonary Artery <7-10 mm
* Subjects with history of recurrent (> 1) pulmonary embolism or deep vein thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten patients receiving hemodialysis treatment will be recruited for the implantation of the CardioMEMS HF System. Five of them will be patients with ESRD caused by polycystic kidney disease or glomerulonephritis with no evidence of cardiovascular disease. The other five will be patients with ESRD and hemodynamical instability during and in between dialysis treatments, defined as ultrafiltration rate minimum of 800 ml/hour and dialysis hypotension.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change of pulmonary artery pressure (PAP) during the dialysis treatment | PAP is recorded every ten minutes during the standard dialysis treatment (4-6h). Measurement is repeated twice a week for one month

SECONDARY OUTCOMES:
Change of pulmonary artery pressure (PAP) in between the dialysis treatment | measurement is made twice a day over the period of one month

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas V Kerola, MD PhD, Principal Investigator — Department of Internal Medicine, Päijät-Häme Central Hospital, Lahti, Finland
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Paijat-Hame Region, Finland

IPD SHARING:
Plan to Share IPD: No